CLINICAL TRIAL: NCT07386704
Title: A Prospective, Single-arm Study of Nimotuzumab Combined With Radiotherapy and Chemotherapy in the Treatment of Unresectable Locally Advanced or Oligometastatic Pancreatic Cancer
Brief Title: Nimotuzumab Combined With Chemoradiotherapy in the Treatment of Unresectable Locally Advanced or Oligometastatic Pancreatic Cancer
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO-A
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer Non-resectable
Keywords: locally advanced; oligometastasis
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab + chemoradiotherapy group (Experimental)
  Interventions: Drug: Nimotuzumab combined with chemoradiotherapy

INTERVENTIONS:
Drug: Nimotuzumab combined with chemoradiotherapy — The patient received treatment with nimotuzumab combined with radiotherapy and chemotherapy. The radiotherapy could be conducted using conventional fractionated radiotherapy or SBRT, and the chemotherapy could be carried out using tegafur or capecitabine.

SUMMARY:
This study is a prospective, single-arm trial, aiming to enroll 30 patients with unresectable locally advanced or oligometastatic pancreatic cancer. The study will evaluate the efficacy and safety of nintedanib combined with radiotherapy and chemotherapy (gemcitabine or capecitabine monotherapy). The primary endpoint of this study is the 1-year local control rate (LCR).

DETAILED DESCRIPTION:
1. Radiotherapy: Conventional fractionated radiotherapy or SBRT can be selected.

1. Conventional Fractionated Radiotherapy: Pancreatic tumor + 5mm PTV 50-60Gy/25 fractions/5W; Pancreatic tumor GTV 60-70Gy/25 fractions/5W; If there are suspected metastatic lymph node regions, prophylactic irradiation of lymph node drainage areas should be performed.
2. Stereotactic Body Radiotherapy (SBRT): Pancreatic tumor + 5mm PTV 30Gy/5 fractions/5 days; Pancreatic tumor GTV 40Gy/5 fractions/5 days.

2. Nintuzumab: Nintuzumab 400mg, intravenous infusion, on day 1, administered once a week (QW). Mix400 mg of nintuzumab injection with 250ml of sodium chloride solution, and the infusion time should be more than 60 minutes. Administer concurrently during radiotherapy and discontinue use after radiotherapy.

3. Chemotherapy (either tegafur or capecitabine, choose one):

1. Tegafur-gimeracil-oteracil (S-1): 80-120mg per day, taken twice a day, from day 1 to day 14, and from day 21 onwards. One treatment cycle consists of 21 days.
2. Capecitabine: 2000mg per square meter per day, taken twice a day, from day 1 to day 14, and from day 21 onwards. One treatment cycle consists of 21 days.

Continue the treatment until the disease progresses or an intolerable toxic reaction occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed by histological or cytological examination as pancreatic adenocarcinoma;
2. Confirmed by imaging as locally advanced or oligometastatic (number of metastatic lesions ≤ 3);
3. Evaluated by the clinical doctor as inoperable or the patient refuses surgery;
4. ECOG PS score 0-1;
5. No radiotherapy has been performed on the upper abdomen before, and no any palliative chemotherapy or other systemic anti-tumor treatment has been received;
6. According to the RECIST 1.1 evaluation criteria, there are measurable lesions;
7. Sufficient organ and bone marrow functions

Exclusion Criteria:

1. Previous history of abdominal radiotherapy.
2. Those with a history of other malignant tumors (excluding cured skin basal cell carcinoma and cervical carcinoma in situ).
3. Those allergic to the drugs or their components used in this protocol.
4. Those with known HIV or syphilis infection, or currently in the active stage of hepatitis (hepatitis B or hepatitis C).
5. Those who have undergone major surgery within 30 days before screening.
6. Those who have used EGFR monoclonal antibody or EGFR-TKI within 30 days before screening.
7. Pregnant or lactating women.
8. Those judged by the investigator to have other reasons unsuitable for participating in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-12-09 (Estimated); Study Completion 2027-12-09 (Estimated)

PRIMARY OUTCOMES:
LCR | The 1-year local control rate (LCR) of patients receiving nivolumab combined with radiotherapy and chemotherapy
  Local Control Rate

SECONDARY OUTCOMES:
OS | The survival rates for 1 year, 2 years, and 5 years
  overall survival
PFS | Every 3 months
  Progression-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiotherapy Oncology, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol